CLINICAL TRIAL: NCT02340143
Title: Assessing Early Behavioral Indicators of Formula Tolerance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mead Johnson Nutrition (Industry)
Collaborators: Baylor College of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: 6025
Record Dates: First submitted 2015-01-06; First posted 2015-01-16 (Estimated); Last update posted 2016-09-14 (Estimated); Status verified 2016-09

CONDITIONS: Tolerance

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Active Comparator): Marketed partially hydrolyzed cow's milk protein infant formula
  Interventions: Other: Control
- Investigational (Experimental): Partially hydrolyzed cow's milk infant formula with a probiotic
  Interventions: Other: Investigational

INTERVENTIONS:
Other: Control — Marketed partially hydrolyzed cow's milk protein infant formula
  Arms: Control
Other: Investigational — Partially hydrolyzed cow's milk protein infant formula with a probiotic
  Arms: Investigational

SUMMARY:
The study is intended to assess the amount of crying and fussiness in infants fed an infant formula containing probiotics.

ELIGIBILITY:
Inclusion Criteria:

* Singleton at birth
* Term infant with birth weight of 2500 g or more
* Crying or fussing for 3 or more hours per day
* Consuming mostly infant formula
* Signed Informed Consent and Protected Health Information authorization

Exclusion Criteria:

* Current use of extensively hydrolyzed or amino acid infant formula
* Planned use of probiotics during the study
* History of underlying metabolic or chronic disease, congenital malformation, or immunocompromised
* Enrollment in another interventional clinical research study

Ages: 14 Days to 28 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 71 (Actual)
Dates: Start 2015-01; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Infant Behavior Diary | 21 Days

SECONDARY OUTCOMES:
Recall of Tolerance Questionnaire | Baseline and Day 21
Body Weight | Baseline and Day 21
Infant Behavior Questionnaire - Revised | Baseline and Day 21
Recall of formula intake at each visit | Baseline, Day 10, and Day 18
Fecal microbiome and Fecal calprotectin | Baseline and Day 21
Medically-confirmed Adverse Events | 21 Days

CONTACTS AND LOCATIONS:
Overall Officials: Carol Lynn Berseth, M.D., Study Director — Mead Johnson Nutrition
Locations (1):
- Children's Nutrition Research Center, Houston, Texas, United States

REFERENCES:
- [Derived] Shulman RJ, Chichlowski M, Orozco FG, Harris CL, Wampler JL, Bokulich NA, Berseth CL. Infant behavioral state and stool microbiome in infants receiving Lactocaseibacillus rhamnosus GG in formula: randomized controlled trial. BMC Pediatr. 2022 Oct 7;22(1):580. doi: 10.1186/s12887-022-03647-x. PMID 36207675